CLINICAL TRIAL: NCT04447651
Title: A Remote-Directed "Virtual" Clinical Trial in Metastatic Solid Tumors to Determine Feasibility of Evaluating Patient Response to Immunotherapy Using Spliceosome Mutational Markers (PRISMM)
Brief Title: Patient Response to Immunotherapy Using Spliceosome Mutational Markers (PRISMM)
Acronym: PRISMM
Status: Active, not recruiting | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Vanderbilt University (Other); Bristol-Myers Squibb (Industry); Avon Breast Health Access Fund (Unknown)
Responsible Party: Sponsor
Other Study IDs: J1940; IRB00186535 (Other: JHM IRB)
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Solid Tumor; SF3B1 Gene Mutation; Spliceosome Mutation; U2AF1 Gene Mutation; SRSF2 Gene Mutation
Keywords: sequencing; metastatic solid tumor; spliceosome mutation; immune checkpoint inhibition; immunotherapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Therapeutics; Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood samples will be collected to:
  * Evaluate whether mutations detected in tumor tissue using various Clinical Laboratory Improvement Amendments (CLIA)-certified next-generation sequencing assays correlate with those found in plasma tumor DNA (ptDNA).
  * To evaluate changes in ptDNA from baseline to 3 months in patients with spliceosome mutations receiving immune checkpoint inhibitors (ICI)
  * To evaluate changes in circulating immune cells (PBMCs) from baseline to 3 months in patients with spliceosome mutations receiving ICI
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with SF3B1, U2AF1 or SRSF2 mutation: Metastatic solid tumor patients that have a SF3B1, U2AF1 or SRSF2 mutation
  Interventions: Other: Recommendation for treatment with immunotherapy

INTERVENTIONS:
Other: Recommendation for treatment with immunotherapy — Patients with a SF3B1, U2AF1 or SRSF2 mutation will be reviewed by the molecular tumor board and treatment recommendations will be given to the patient's treating oncologist.

SUMMARY:
This study is being done to see if patients with metastatic solid tumors (hematologic malignancies and lymphoma excluded) who have a specific genetic mutation in patients' tumor (the SF3B1, U2AF1 or SRSF2 mutation), are more likely to respond to immunotherapy agents that are now commercially available.

DETAILED DESCRIPTION:
This is a non-therapeutic study, meaning that while Johns Hopkins is providing a treatment recommendation based on participants' genetic information, participants and participants' oncologist will decide ultimately what to do, and participants' oncologist will monitor participants' day to day care while on therapy. Participation involves allowing the investigators access to participants' sequencing report and medical records, providing a blood sample (about 8 tablespoons) at baseline and possibly again after three months, and answering questionnaires. If participants join the study, a panel of experts (Johns Hopkins Molecular Tumor Board) will review participants' genetic information participants entered and make a determination regarding treatment recommendation. Blood will be collected at baseline irrespective of what treatment is recommended. If immunotherapy is recommended, the investigators may collect blood again at 3 months. Participants and participants' oncologist will ultimately decide if participants proceed with the recommend treatment or not; the recommendation made from Johns Hopkins is not binding in any way. Participants' oncologist will continue with usual care according to standard practices while participants are on therapy. The investigators will get health information and conduct questionnaires with participants and participants' oncologist to assess how participants are doing on therapy. The main risks are the discomforts of the blood draw (which are expected to be minor and not last), boredom from completing questionnaires and the risk that information may become known to people outside of the study. Participants may or may not benefit directly from being in the study and there is no payment for participation.

ELIGIBILITY:
Inclusion Criteria:

* Performance status eligible for immune checkpoint blockade as determined by local physician
* Able to demonstrate histologically proven locally advanced or metastatic solid tumors (hematologic malignancies and lymphoma excluded)
* genomic testing demonstrating a spliceosome mutation (SF3B1, U2AF1 or SRSF2)

Exclusion Criteria:

* Local physician determines has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Local physician determines the patient has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic solid tumor patients with a SF3B1,U2AF1 or SRSF2 mutation.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of study as assessed by completion of study accrual within study time frame | 2 years
  To evaluate the feasibility of conducting a prospective study using online recruitment tools to involve patients and physicians who are not usually served by clinical trials. Measured by enrolling 60 patients over 2 years.
Feasibility of study as assessed by physician responses | 1 year
  To evaluate the feasibility of conducting a prospective study using online recruitment tools to involve patients and physicians who are not usually served by clinical trials. Measured by obtaining responses from 80 percent of physicians within 1 year of enrollment.
Feasibility of case review as assessed by time to issuance of recommendations | 4 weeks from consent
  To evaluate the feasibility of real-time case review by a centralized specialized cancer tumor board to assist in therapeutic decision making. Measured by time (days) to issuance of recommendations within 4 weeks from consent for at least 80 percent of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Santa-Maria, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States